Lifebox Project IRAS No: 211895



Great Ormond Street London WC1N 3JH T: +44 (0)20 7405 9200

## Development of a robust and reliable pulse oximeter for use by frontline healthcare providers caring for children with pneumonia in low-income countries

**CONSENT FORM** 

This study (Project ID: 15HC31) has been given favourable review for conduct in the NHS by: XXXX Research Ethics Committee on date YYYY

| Naı | mα | Λf | Ch | ١ĭ١ | | ۰ |
|------|-----|----|----|-----|---|---|
| ıvaı | 116 | Οī | CI | Ш | u | • |

Please initial all boxes

| 1. | firm that I have read and understand the information sheet dated XXX (version 1.0) for the above. I have had the opportunity to consider the information and ask questions and I have had my ions answered satisfactorily. |
|---|---|
| 2. | I understand that my child's participation is voluntary and that I am free to withdraw consent for my child to participate at any time without giving any reason, without my child's medical care or legal rights being affected. |
| 3. | I understand that information provided for this study will be treated as strictly confidential and handled in accordance with the Data Protection Act 1998. I am assured that no personal identifying information will be kept which could link my child to any data recorded. |
| 4. | I understand that data collected during the study may be looked at by individuals from Great Ormond Street Hospital, or from regulatory authorities. I give permission for these individuals to have access to my child's records. |
| 5. | I give permission for my child to take part in this study |
| Nar | ne of parent/guardian Date Signature |

You will be given a copy of this information sheet and signed consent form for your records.

Thank you for your time.

Signature

Date

Parent consent form

Name of person taking consent

Date of issue: 24<sup>th</sup> October 2016 Consent form version number: v1